CLINICAL TRIAL: NCT05752370
Title: Improving Post-hospitalization Outcomes of Respiratory Patients With Exertional Hypoxemia by Early Pulmonary Rehabilitation Using High Flow Nasal Oxygen- a Pilot Randomized Controlled Trial.
Brief Title: Improving Outcomes of Respiratory Patients With Exertional Hypoxemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/2605
Record Dates: First submitted 2023-02-13; First posted 2023-03-02 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Pulmonary Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow oxygen (Experimental): High flow nasal oxygen
  Interventions: Device: High flow oxygen
- Usual care (Active Comparator): room air or normal flow oxygen
  Interventions: Other: Usual care

INTERVENTIONS:
Device: High flow oxygen — Use of HFO
  Arms: High flow oxygen
Other: Usual care — Room air or normal flow oxygen
  Arms: Usual care

SUMMARY:
The primary aim of this pilot randomized controlled trial is to determine feasibility of the proposed pulmonary rehabilitation intervention.

DETAILED DESCRIPTION:
In this pilot randomized controlled trial, our primary aim is to determine feasibility of the proposed intervention.

ELIGIBILITY:
Inclusion Criteria:

* 21 years and above
* Presence of exertional hypoxemia during 1-minute sit-to-stand test
* diagnosis of acute COPD exacerbation or Covid-19 pneumonia or exacerbation of bronchiectasis or exacerbation of interstitial lung disease
* physically fit to participate in exercise therapy as determined by both the patient's physician and physiotherapist

Exclusion Criteria:

* uncontrolled severe medical conditions
* currently enrolled in a pulmonary rehabilitation trial
* unsuitable for randomization as determined by the patient's physician

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in 1-minute sit to stand test | 1 month
  maximum number of sit to stand cycles in 1 minute

SECONDARY OUTCOMES:
Changes in 30-second sit to stand test | 1 month, 3 month
  maximum number of sit to stand cycles in 30 seconds
Changes in respiratory symptoms | 1 month, 3 months
  Modified Medical Research Council Dyspnea Scale. The scale ranges from 0 to 4 with a higher score indicating increasing breathlessness
Changes in mood | 1 month, 3 month
  Hospital Anxiety Depression Scale. The scale ranges from 0 to 21, A total subscale score of >8 points indicates considerable symptoms of anxiety or depression.
changes in quality of life | 1 month, 3 month
  EQ-5D-5L
Changes in lung function | 1 month, 3 month
  Forced expiratory volume in 1 sec
Changes in lung function | 1 month, 3 month
  forced vital capacity
Proportion of patients who still have exertional hypoxemia | 1 month, 3 month
  Comparing the proportion of patients who still have exertional hypoxemia
Adherence rates | 3 week
  Comparing the adherence rates between the 2 study arms
Changes in 1-minute sit to stand test | 3 month
  maximum number of sit to stand cycles in 1 minute

OTHER OUTCOMES:
Qualitative interview | Upon completion of study, or when patients end participation in the study
  Qualitative interviews will also be conducted to obtain patient perspectives of the interventions in the study

CONTACTS AND LOCATIONS:
Overall Officials: Yingjuan Mok, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No